CLINICAL TRIAL: NCT04212481
Title: Randomized Controlled Trial of the Comparison of Uniport VATS and Non- Uniport VATS for Lung Cancer
Brief Title: RCT of Uniport VATS for Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uniport VATS ZYP1
Record Dates: First submitted 2019-12-21; First posted 2019-12-27 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Single-port Video-assisted Thoracoscopic Surgery
Keywords: Non Small Cell Lung Cancer; Perioperative Efficacy; multi-port
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single port group (Experimental): Uniport video-assisted thoracoscopic surgery for NSCLC
  Interventions: Procedure: uniport video-assisted thoracoscopic surgery
- two ports group (Active Comparator): video-assisted thoracoscopic surgery for NSCLC using two ports
  Interventions: Procedure: two ports video-assisted thoracoscopic surgery
- three ports group (Active Comparator): video-assisted thoracoscopic surgery for NSCLC using three ports
  Interventions: Procedure: three ports video-assisted thoracoscopic surgery

INTERVENTIONS:
Procedure: uniport video-assisted thoracoscopic surgery — video-assisted thoracoscopic surgery for NSCLC using single port or two ports or three ports
  Arms: single port group
Procedure: two ports video-assisted thoracoscopic surgery — video-assisted thoracoscopic surgery for NSCLC using two ports
  Arms: two ports group
Procedure: three ports video-assisted thoracoscopic surgery — video-assisted thoracoscopic surgery for NSCLC using three ports
  Arms: three ports group

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) has been widely used for non-small cell lung cancer (NSCLC) for nearly two decades. Usually, it was applied through three ports with at least one drainage after surgery, which often lead to acute chest pain. Therefore, fewer, smaller ports, and wider intercostal space for surgery has been required.

Uniport VATS became a feasible option with the development of surgical techniques and instruments, with potentially less postoperative pain and shorter hospital stays. However, there may be some complications, or with a longer time of operation, even more difficult in lymph nodes resection during learning curve.

In our study, a Randomized Controlled Trial was designed to study the operation time, perioperative blood loss, conversion rate, duration of postoperative drainage, length of hospital stay, visual analogue score of postoperative pain, complications, and survival.

ELIGIBILITY:
Inclusion Criteria:

patients with cT1-3N0-1M0 NSCLC; good cardiopulmonary function; prepared to undergo radical resection;

Exclusion Criteria:

patients with N3 or M1 NSCLC; poor cardiopulmonary function; not be prepared to undergo radical resection;

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-12-25 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
operative time | 1 day
  operative time in minutes
perioperative blood loss | 1 day
  perioperative blood loss in milliliter
conversion rate | 1 day
  conversion rate in proportion
duration of postoperative drainage | within 5-7 days
  duration of postoperative drainage in days
length of hospital stay | within 5-7 days
  length of hospital stay in days
visual analogue score of postoperative pain | within 5-7 days
  score
complications | up to 3 months
  complications in rate

SECONDARY OUTCOMES:
overall survival | up to 5 years
  overall survival in rate
progression- free survival | up to 5 years
  progression- free survival in rate

CONTACTS AND LOCATIONS:
Overall Officials: Xiaogang Zhao, Doctor, Study Director — The Second Hospital of Shandong University
Locations (1):
- The Second Hospital of Shandong University, Jinan, Shandong, China